CLINICAL TRIAL: NCT02588560
Title: Serial Viral Load Changes and Hepatotoxicity in Lymphoma Patients With Hepatitis C Antibody After Chemotherapy Treatment: A Prospective Multicenter Observational Study and Long-term Retrospective Analysis
Brief Title: Viral Load Changes in Lymphoma Patients With HCV Infection After Chemotherapy
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 103-7486B
Record Dates: First submitted 2015-10-16; First posted 2015-10-28 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-08

CONDITIONS: Lymphoma; Hepatitis C Antibodies; Drug Therapy
Keywords: lymphoma, hepatitis C virus, chemotherapy
MeSH Terms: conditions — Lymphoma; Hepatitis C

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood mononuclear cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HCV lymphoma patients with chemotherapy: Lymphoma patients who are positive for anti-HCV and are planning to receive chemotherapy for lymphoma

SUMMARY:
In last few years, most researches about hepatic complication after chemotherapy focused on hepatitis B virus (HBV). With adequate prophylaxis and monitor, HBV-related hepatitis flares can be prevented. In contrast, cancer patients with hepatitis C virus (HCV) infection are traditionally considered as relative safe to receive chemotherapy. However, two large retrospective studies recently showed that severe hepatitis could develop in 14-27% lymphoma patients with chronic HCV infection, including 3-4% hepatic failure. The risk factors to predict severe hepatitis are pre-treatment elevated ALT level and liver cirrhosis. Due to the lack of prospective studies, the dynamic changes of serum HCV RNA levels and the association of hepatitis are still unclear.

Some epidemiologic studies demonstrated an association between HCV infection and B-cell lymphoma. Diffuse large B-cell lymphoma (DLBCL) is the most common lymphoma and several reports showed higher prevalence of HCV infection among DLBCL patients than the controls. HCV infected DLBCL patients are reported to have distinct clinical characteristics, such as older, more with elevated LDH levels, and more with extra-nodal involvement. Regarding the impact of HCV infection on prognosis, the results are conflicting. Taiwan is an endemic area of HCV but there are limited reports addressing the clinical characteristics and prognosis in this unique population.

Therefore, the investigators initiate a prospective, multi-center observational study to clarify the dynamic association between serum HCV RNA levels and hepatitis in HCV-infected lymphoma patients treated with chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed histologically proven malignant lymphoma
2. Eligible subjects must be positive for anti-HCV Ab
3. Age ≥ 20 years
4. Planned to receive chemotherapy
5. No recent chemotherapy and radiotherapy in the past one year. Pre-enrollment steroids for symptomatic relief are allowed but less than equivalent dose to prednisolone total 140 mg
6. Left expectancy ≥ 3 months
7. Signed informed consent
8. ECOG 0-2

Exclusion Criteria:

1. Patients not willing to receive chemotherapy
2. Chronic hepatitis B infection (positive for HBsAg), but those with resolved HBV infection (positive for anti-HBc and negative for HBsAg) are allowed
3. Other major systemic diseases, such as active infection, significant cardiac disease, neurologic deficit or psychiatric disorders, that the investigators consider to be at significant risk
4. Known human immunodeficiency virus (HIV) infection
5. Pregnant or breast-feeding woman

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lymphoma patient plus hepatitis C
Sampling Method: Non-Probability Sample
Enrollment: 38 (Estimated)
Dates: Start 2015-09; Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Increasing HCV RNA Level and Developing Hepatitis after Chemotherapy | one year
Number of Participants with Detectable Viremia and Developing Hepatitis after Chemotherapy | one year
Interval (months) between Peak HCV RNA Level and Hepatitis | one year
Increase (log) of HCV Viral Load between Baseline and after Chemotherapy | one year

SECONDARY OUTCOMES:
Number of Participants with Hepatitis after Chemotherapy | one year
  Hepatitis is defined as ALT level > 2.5X ULN
Number of Participants with Severe Hepatitis after Chemotherapy | one year
  Severe hepatitis is defined as ALT level > 5X ULN or Bilirubin level > 3.0X ULN
Number of Participants with Chemotherapy Interruption due to Hepatotoxicity | one year
Number of Participants with Early Stop of Chemotherapy due to Hepatotoxicity | one year